CLINICAL TRIAL: NCT05244707
Title: The Effects of a Mediterranean Style Diet in Heart Disease Patients Running a Cardiac Rehabilitation Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Nova de Lisboa (Other)
Collaborators: Hospital de Santa Marta - Centro Hospitalar Universitário, Lisboa Central (CHULC), Portugal (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NutriReHeart
Record Dates: First submitted 2022-02-07; First posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Acute Myocardial Infarction With ST Elevation
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean style diet (Experimental): Mediterranean style diet.
  Interventions: Behavioral: Mediterranean style diet
- Standard of care (Active Comparator): Standard of care.
  Interventions: Behavioral: Standard of care

INTERVENTIONS:
Behavioral: Mediterranean style diet — The intervention will consist of an intensive food and nutrition intervention program to improve adherence to the Mediterranean dietary pattern. In addition to individual and face-to-face nutrition consultations, other strategies will be used, such as telephone contacts, short text messages, consultation support tools, podcasts, short open access videos, nutrition workshops and nutrition sessions for caregivers of participants in the study.
  Arms: Mediterranean style diet
Behavioral: Standard of care — The usual care group will only have access to face-to-face and individual nutrition consultations in order to improve adherence to the Mediterranean dietary pattern.
  Arms: Standard of care

SUMMARY:
Nutrition is capable of altering the cardiovascular health of the general population. However, the ideal food and nutritional interventions for the secondary prevention of cardiovascular brain disease and for cardiac rehabilitation are still far from being defined, given the lack of scientific evidence in this specific population of individuals with atherosclerotic disease. This work aims to demonstrate that an intensive program will improve cardiovascular risk predictor parameters, such as high systolic blood pressure, altered lipid and glucose profile, used in the SMART Risk Score tool. In this 12-week clinical study with two arms running in parallel, individuals referred to a cardiac rehabilitation program will receive either an intensive food and nutrition intervention program with nutrition consultations, in which the adoption of the Mediterranean diet is promoted, with contacts telephone calls, short text messages, consultation support tools, podcasts, free access short videos, culinary medicine sessions and nutrition "workshops", or the standard of care program recommended in the Nutritional Support Protocol of the Cardiac Rehabilitation Program. At the beginning of the study, at 4 weeks, at 8 weeks and at 12 weeks, blood and urine samples will be collected, body composition, blood pressure, adherence to the Mediterranean dietary pattern will be assessed, by applying the PREDIMED questionnaire and the dietary intake of 24h previous. The quality of life of individuals will be assessed by the EQ-5D-5L questionnaire at the beginning and at the end of the study. It is expected that the increased intensity and support from the intensive program will have a significant impact on the various metabolic and inflammatory markers predictive of cardiovascular risk and that these observed changes will result in a decreased 10-year risk of developing acute myocardial infarction, stroke or vascular death. On the other hand, the intervention is intended to improve quality of life, improve weight control and assess the impact it has on adherence to the Mediterranean dietary pattern.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with ST-segment elevation acute myocardial infarction undergoing primary angioplasty;
* Ages 30-90 years;
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Subjects with heart failure (LVEF <50% or NT_proBNP> 125 ng / mL) on admission;
* Subjects with renal failure (GFR <50 or 60 ml / min / 1.73m²);
* Subjects requiring internment;
* Subjects who present any other condition that may interfere with adherence to the study protocol.

  * Subjects who attract to be accompanied by another nutritionist;
  * Subjects who have a specific dietary pattern or who take vitamin and/or mineral supplements;
  * Subjects unable to give consent.

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in SMART Risk Score | baseline to 12 weeks
  Difference between the intervention and control group in the change in SMART Risk Score from baseline to the end of follow-up.

SECONDARY OUTCOMES:
Self-reported quality of life | baseline to 12 weeks
  Difference between the intervention and control group in the EQ-5D-5L questionnaire from baseline to the end of follow-up.
Adherence to the Mediterranean dietary pattern | baseline, 4 weeks, 8 weeks and 12 weeks
  Difference between the intervention and control group in MEDAS questionnaire from baseline to 4 weeks, 8 weeks and 12 weeks.
Change in weight | baseline to 12 weeks
  Difference between the intervention and control group in the change of weight (kg) from baseline to 12 weeks.
Change in body fat | baseline to 12 weeks
  Difference between the intervention and control group in the change of body fat (%) from baseline to 12 weeks.
Change in fat free mass | baseline to 12 weeks
  Difference between the intervention and control group in the change of fat free mass (kg) from baseline to 12 weeks.
Change in total body water | baseline to 12 weeks
  Difference between the intervention and control group in the change of total body water (kg) from baseline to 12 weeks.
Change in systolic blood pressure | baseline, 4 weeks, 8 weeks and 12 weeks
  Difference between the intervention and control group in the change of systolic blood pressure from baseline to 4 weeks, 8 weeks and 12 weeks.
Change in diastolic blood pressure | baseline, 4 weeks, 8 weeks and 12 weeks
  Difference between the intervention and control group in the change of diastolic blood pressure from baseline to 4 weeks, 8 weeks and 12 weeks.
Change of insulin | baseline, 4 weeks, 8 weeks and 12 weeks
  Difference between the intervention and control group in the change of insulin from baseline to 4 weeks, 8 weeks and 12 weeks.
Change of fasting blood glucose | baseline, 4 weeks, 8 weeks and 12 weeks
  Difference between the intervention and control group in the change of fasting blood glucose from baseline to 4 weeks, 8 weeks and 12 weeks.
Change of glycosylated hemoglobin (HbA1c) | baseline, 4 weeks, 8 weeks and 12 weeks
  Difference between the intervention and control group in the change of glycosylated hemoglobin (HbA1c) from baseline to 4 weeks, 8 weeks and 12 weeks.
Change of type 1 insulin-like growth factor (IGF-1) | baseline, 4 weeks, 8 weeks and 12 weeks
  Difference between the intervention and control group in the change of type 1 insulin-like growth factor (IGF-1) from baseline to 4 weeks, 8 weeks and 12 weeks.
Change of LDL cholesterol | baseline, 4 weeks, 8 weeks and 12 weeks
  Difference between the intervention and control group in the change of LDL- cholesterol from baseline to 4 weeks, 8 weeks and 12 weeks.
Change of HDL cholesterol | baseline, 4 weeks, 8 weeks and 12 weeks
  Difference between the intervention and control group in the change of HDL- cholesterol from baseline to 4 weeks, 8 weeks and 12 weeks.
Change of triglycerides | baseline, 4 weeks, 8 weeks and 12 weeks
  Difference between the intervention and control group in the change of triglycerides from baseline to 4 weeks, 8 weeks and 12 weeks.
Change of apolipoprotein B | baseline, 4 weeks, 8 weeks and 12 weeks
  Difference between the intervention and control group in the change of apolipoprotein B from baseline to 4 weeks, 8 weeks and 12 weeks.
Change of apolipoprotein A1 | baseline, 4 weeks, 8 weeks and 12 weeks
  Difference between the intervention and control group in the change of apolipoprotein A1 from baseline to 4 weeks, 8 weeks and 12 weeks.
Change of liporprotein(a) | baseline, 4 weeks, 8 weeks and 12 weeks
  Difference between the intervention and control group in the change of liporprotein(a) from baseline to 4 weeks, 8 weeks and 12 weeks.
Change of high sensitivity C-reactive protein | baseline, 4 weeks, 8 weeks and 12 weeks
  Difference between the intervention and control group in the change of high sensitivity C-reactive protein from baseline to 4 weeks, 8 weeks and 12 weeks.
change of myeloperoxidase | baseline, 4 weeks, 8 weeks and 12 weeks
  Difference between the intervention and control group in the change of myeloperoxidase from baseline to 4 weeks, 8 weeks and 12 weeks.
Change of interleukin 1 | baseline, 4 weeks, 8 weeks and 12 weeks
  Difference between the intervention and control group in the change of interleukin 1 from baseline to 4 weeks, 8 weeks and 12 weeks.
Change of interleukin 6 | baseline, 4 weeks, 8 weeks and 12 weeks
  Difference between the intervention and control group in the change of interleukin 6 from baseline to 4 weeks, 8 weeks and 12 weeks.
Change of tumor necrosis factor alpha (TNF-α) | baseline, 4 weeks, 8 weeks and 12 weeks
  Difference between the intervention and control group in the change of tumor necrosis factor alpha (TNF-α) from baseline to 4 weeks, 8 weeks and 12 weeks.
Change of trimethylamine N-oxide (TMAO) | baseline, 4 weeks, 8 weeks and 12 weeks
  Difference between the intervention and control group in the change of trimethylamine N-oxide (TMAO) from baseline to 4 weeks, 8 weeks and 12 weeks.
Change of L-carnitine | baseline, 4 weeks, 8 weeks and 12 weeks
  Difference between the intervention and control group in the change of L-carnitine from baseline to 4 weeks, 8 weeks and 12 weeks.
Change of urinary hydroxytyrosol | baseline, 4 weeks, 8 weeks and 12 weeks
  Difference between the intervention and control group in the change of urinary hydroxytyrosol from baseline to 4 weeks, 8 weeks and 12 weeks.
Change of plasma proportion of alpha linolenic acid | baseline, 4 weeks, 8 weeks and 12 weeks
  Difference between the intervention and control group in the change of plasma proportion of alpha linolenic acid from baseline to 4 weeks, 8 weeks and 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Rio, MD, Principal Investigator — Hospital de Santa Marta - Centro Hospitalar Universitário | Lisboa Central (CHULC); Conceição Calhau, PhD, Principal Investigator — NOVA Medical School | Faculdade de Ciências Médicas da Universidade NOVA de Lisboa; André Moreira-Rosário, PhD, Study Director — NOVA Medical School | Faculdade de Ciências Médicas da Universidade NOVA de Lisboa; Júlio C Rocha, PhD, Study Director — NOVA Medical School | Faculdade de Ciências Médicas da Universidade NOVA de Lisboa; Diana Teixeira, PhD, Study Director — NOVA Medical School | Faculdade de Ciências Médicas da Universidade NOVA de Lisboa